CLINICAL TRIAL: NCT03368456
Title: Preventing HIV/STI in Urban Adolescents Via an mHealth Primary Care Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David Cordova, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00158089; Previous HUM00118704 (Other: University of Michigan IRB)
Record Dates: First submitted 2017-11-20; First posted 2017-12-11 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: HIV/AIDS and Infections; Drug Abuse; Adolescent Behavior; Drug Usage
Keywords: mhealth; preventive intervention; primary health care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Substance-Related Disorders; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: To test the preliminary efficacy of S4E, we will conduct a Stage I RCT and use a mixed between/within-subjects design with two levels of intervention (S4E and Usual Care) as the between-subjects factor and three repeated measures assessments (Baseline, 3-, and 6-months post-Baseline) as the within-subjects factor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S4E App Intervention (Experimental): Participants in the S4E condition will first receive the intervention in the waiting area via iPads provided for them. Content includes the theoretically driven components of Storytelling for Empowerment: (a) Storytelling scenarios, (b) drug use and HIV/STI knowledge development, (c) interactive activities, (d) increasing self-efficacy to prevent/reduce sexual risk and drug use behaviors, and increase HIV/STI testing, (e) clinician-youth communication, and (f) highlighting prevention principles
  Interventions: Behavioral: S4E
- Usual Care Condition (Placebo Comparator): Participants in Usual Care (i.e., Control Condition) will not receive the S4E intervention. The Clinic's usual care includes a standard risk behaviors intake form, pamphlets highlighting resources, and reproductive and healthcare services.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: S4E — S4E application was developed in collaboration with youth in Southeast Michigan. S4E aims to prevent and reduce HIV/STI risk behaviors, including drug use and sexual risk behaviors, and increase HIV/STI testing among youth. Content produced for the application is based on scientific prevention principles in conjunction with youth input. To date, we have developed modules focused on youth alcohol & drug use, HIV & STIs and a forthcoming module on tobacco prevention and cessation.
  Arms: S4E App Intervention
Behavioral: Usual Care — Participants in Usual Care (i.e., Control Condition) will not receive the S4E intervention from the study staff. The Clinic's usual care includes a standard risk behaviors intake form, pamphlets highlighting resources, and reproductive and healthcare services.
  Arms: Usual Care Condition

SUMMARY:
The study evaluates the preliminary efficacy of an innovative mobile-health (mHealth) intervention (hereon referred to as S4E) to improve human immunodeficiency virus and sexually transmitted infection testing and reduce HIV/STI risk behaviors in a clinic sample (n=100) of at-risk youth ages 14-21 living in Southeast Michigan. A Stage I randomized control trial will be conducted to examine the preliminary efficacy of S4E, relative to Usual Care (UC), over a period of six months.

DETAILED DESCRIPTION:
HIV/STI and drug abuse remain significant public health priorities in the US and youth are disproportionately affected. Youth between the ages of 15 - 24 constitute 25% of the sexually experienced population, yet account for 46% and 50% of HIV infections and new STIs, respectively. National surveillance data indicate that youth disproportionately engage in HIV/STI risk behaviors, including condomless sex and licit and illicit drug use, which increase their risk for HIV/STI infection. Despite the disproportionately high rates of HIV/STI infection and risk behaviors in youth, fewer than 14% report having ever been tested for HIV and many are not routinely screened for asymptomatic STIs as recommended by the Center for Disease Control. In Southeast Michigan, HIV/STI are disproportionately high. To address these significant public health concerns, a mobile-health (mHealth) intervention was developed for health clinic settings. The proposed research aims to develop a cross-platform and universal version of S4E. The cross-platform and universal version of S4E will be compatible with both IOS and Android operating systems, and multiple mobile devices, aimed at providing adolescents with ongoing access to the intervention once they leave the clinic. The proposed research will also evaluate the preliminary efficacy of S4E to improve HIV/STI testing and reduce HIV/STI risk behaviors in a clinic sample (n=100) of at-risk youth ages 14-21 living in Southeast Michigan by conducting a Stage I RCT to examine the preliminary efficacy of S4E, relative to Usual Care, among a sample of 100 at-risk youth over six months.

ELIGIBILITY:
Inclusion Criteria:

* Female or male youth 14-21 years of age
* Sexually active
* Live in Southeast Michigan
* Have access to a smartphone or tablet
* Youth must see an enrolled clinician to participate in the study.

Exclusion Criteria:

* Report of prior psychiatric hospitalization by adolescent
* Visible cognitive impairment due to drug use
* Adolescent reports (tentative or firm) plans to move out of the Southeast Michigan area during the study

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Change in Adolescent HIV Testing | baseline, 3 and 6 month post-baseline
  Post-intervention, we will assess whether youths requested to receive HIV testing at the clinic, and at 3 and 6 months post-baseline (yes/no).

SECONDARY OUTCOMES:
Change in condomless sex behaviors | 3 and 6 month post-baseline
  Adolescent unsafe sexual behavior will be measured (time points 1-3) using items extracted from Jemmott, Jemmott, and Fong's Sexual Behavior instrument. This gated instrument will assess the adolescent's past 90-day condom use, number of sexual partners, and contraceptive use (non-condom).
Change in drug use behaviors | baseline, 3 and 6 month post-baseline
  Licit and illicit drug use behaviors will be assessed (time points 1-3) using items from the Monitoring the Future Study. Youth will be asked whether or not they have used licit or illicit drugs in their lifetime and the past 90 days. Youth who report "Yes" to past 90-day sex will be asked to report the frequency of drug use before sex. These measures have been used in our formative research.

OTHER OUTCOMES:
Change in Clinician-Youth Communication | baseline, 3 and 6 month post-baseline
  Completed by both the clinician (α =.70) and youth (α =.69), clinician-youth communication will be assessed (time points 1-3) using items adapted from the Matched Pair Instrument (19 items; MPI). MPI assesses process and content of communication, including verbal and action-related behaviors performed by clinicians. Responses range from "1=strongly disagree," to "5=strongly agree," on a five-point Likert scale. A sample statement for clinicians and youths is, "Encouraged the patient/me to express his or her/my thoughts concerning drug use behaviors."
Youth Self-Efficacy | baseline, 3 and 6 month post-baseline
  Youth's self-efficacy will be assessed (time points 1-3) using two scales, including the Condom Self-Efficacy Scale (19 items, α =.85), and Drug Use Resistance Self-Efficacy (24 items, α =.98). Responses range from "1=not sure at all," to "4=definitely sure," on a four-point Likert scale. A sample question for the youth is, "How sure are you that you can refuse if a friend offers you marijuana at a party and you do not want it?"

CONTACTS AND LOCATIONS:
Overall Officials: David Cordova, PhD, Principal Investigator — University of Michigan
Locations (1):
- Corner Health Center, Ypsilanti, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordova D, Alers-Rojas F, Lua FM, Bauermeister J, Nurenberg R, Ovadje L, Fessler K, Delva J, Salas-Wright CP, Council YL. The Usability and Acceptability of an Adolescent mHealth HIV/STI and Drug Abuse Preventive Intervention in Primary Care. Behav Med. 2018 Jan-Mar;44(1):36-47. doi: 10.1080/08964289.2016.1189396. Epub 2016 Jul 15. PMID 27223646
- [Background] Cordova D, Bauermeister JA, Fessler K, Delva J, Nelson A, Nurenberg R, Mendoza Lua F, Alers-Rojas F, Salas-Wright CP; Youth Leadership Council. A Community-Engaged Approach to Developing an mHealth HIV/STI and Drug Abuse Preventive Intervention for Primary Care: A Qualitative Study. JMIR Mhealth Uhealth. 2015 Dec 18;3(4):e106. doi: 10.2196/mhealth.4620. PMID 26685288
- [Derived] Cordova D, Bauermeister JA, Warner S; Youth Leadership Council; Wells P, MacLeod J, Neilands TB, Mendoza Lua F, Delva J, Fessler KB, Smith V Jr, Khreizat S, Boyer C. Efficacy of a Digital Health Preventive Intervention for Adolescents With HIV or Sexually Transmitted Infections and Substance Use Disorder: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 19;13:e47216. doi: 10.2196/47216. PMID 38373025

DOCUMENTS (1):
  • Informed Consent Form (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03368456/ICF_000.pdf